CLINICAL TRIAL: NCT06938113
Title: Efficacy and Safety of Flexible Ureteroscope Combined With Flexible Vacuum-assisted Sheath for Intelligent Pressure Control in the Treatment of Kidney Stones
Brief Title: Ureteroscopy Combined With Negative Pressure Sheath Treatment of Kidney Stones
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NP-URL
Record Dates: First submitted 2025-03-26; First posted 2025-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The removal rate, complication risk and operation time of ureteral soft scope combined with negative pressure suction sheath therapy for patients with high-load kidney stones (2-3cm) are still controversial. Therefore, the safety and effectiveness of flexible ureteroscope combined with negative pressure suction sheath in treating patients with high-load kidney stones is unknown. This study will help to solve the problems, provide a more scientific treatment strategy for clinical practice, and promote the application of negative pressure aspiration technology in the field of flexible ureteroscopy lithotripsy, providing new means and ideas for individualized treatment.

DETAILED DESCRIPTION:
The patients enrolled in the group should complete the routine clinical diagnosis and treatment before the operation, including non-contrast CT scan of the urinary system (before surgery), urine routine, urine culture, etc. The postoperative follow-up mainly includes complications after the operation, the time of removing the D-J tube, the time of removing the urinary catheter, urine routine, urine culture, etc. The blood routine, blood chemistry, etc. should be reexamined in the outpatient department one month (4 weeks) after the operation.Patients underwent low-dose CT (DLP:0.45 mGy·cm) scans on the first day and one month after surgery.

During the operation, we will collect some data, including the time when invasive procedures start, the total operation time, the renal pelvis pressure, laser power, and total laser energy; we will also keep a backup of the operation video.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with kidney stones with a diameter of 2-3cm by computed tomography;
2. Age > 18 years old;
3. The anatomical structure of the kidney is normal, without deformity;
4. No serious heart and lung disease (ASA grade I-III)
5. Through preoperative communication, patients and their family members indicated that they were fully aware of the condition and the choice of treatment plan, and signed informed consent and informed choice notification;

Exclusion Criteria:

1. Simultaneous operation is required for ipsilateral ureteral calculi or contralateral upper or lower urinary calculi.
2. Severe coagulation dysfunction;
3. Patients who do not sign informed consent and cannot cooperate with the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age range from 18 to 75 years old; Patients undergoing flexible ureteroscopy lithotripsy in our hospital due to high-load kidney stones(2-3cm); All enrolled patients received informed consent and signed informed consent before operation.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Stone removal rate 1 month after surgery | From enrollment to 1 month after surgery

SECONDARY OUTCOMES:
Immediate stone free rate | From enrollment to 1 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China